CLINICAL TRIAL: NCT02864420
Title: Hospitalization at Home Pilot: The Acute Care Home Hospital Program for Adults
Brief Title: Hospitalization at Home: The Acute Care Home Hospital Program for Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Partners HealthCare (Other); Smiths Medical, ASD, Inc. (Industry); Vital Connect, Inc. (Unknown)
Responsible Party: Principal Investigator, Jeffrey L. Schnipper, MD.,MPH., Associate Physician, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001337
Record Dates: First submitted 2016-08-03; First posted 2016-08-12 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Pneumonia; Heart Failure; Cellulitis; Urinary Tract Infections
Keywords: home hospital; acute care home; care redesign; delivery innovation; heart failure; pneumonia; cellulitis; urinary tract infections
MeSH Terms: conditions — Pneumonia; Heart Failure; Cellulitis; Urinary Tract Infections | interventions — Length of Stay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inpatient hospitalization (Active Comparator): Control / usual care arm. Patients are admitted per usual to an inpatient service. Patients' medical records will be closely monitored. Patients will wear a vitals and activity monitor whose data is used only retrospectively. On discharge and 30 days after discharge, they will be interviewed regarding their hospitalization and health.
  Interventions: Other: Inpatient Hospitalization
- Home hospitalization (Experimental): Intervention arm. Patients will return home after triage, diagnosis, and the beginning of treatment in the emergency department with a set of specialized patient-tailored services (listed above). On discharge and 30 days after discharge, they will be interviewed regarding their hospitalization and health.
  Interventions: Other: Home hospitalization

INTERVENTIONS:
Other: Home hospitalization
  Arms: Home hospitalization
Other: Inpatient Hospitalization
  Arms: Inpatient hospitalization

SUMMARY:
The investigators propose a home hospital model of care that substitutes for treatment in an acute care hospital. Limited studies of the home hospital model have demonstrated that a sizeable proportion of acute care can be delivered in the home with equal quality and safety, reduced cost, and improved patient experience.

DETAILED DESCRIPTION:
Hospitals are the standard of care for acute illness in the United States, but hospital care is expensive and often unsafe, especially for older individuals. While admitted, 20% suffer delirium, over 5% contract hospital-acquired infections, and most lose functional status that is never regained. Timely access to inpatient care is poor: many hospital wards are typically over 100% capacity, and emergency department waits can be protracted. Moreover, hospital care is increasingly costly: many internal medicine admissions have a negative margin (i.e., expenditures exceed hospital revenues) and incur patient debt.

The investigators propose a home hospital model of care that substitutes for treatment in an acute care hospital. Studies of the home hospital model have demonstrated that a sizeable proportion of acute care can be delivered in the home with equal quality and safety, 20% reduced cost, and 20% improved patient experience. While this is the standard of care in several developed countries, only 2 non-randomized demonstration projects have been conducted in the United States, each with highly local needs. Taken together, home hospital evidence is promising but falls short due to non-robust experimental design, failure to implement modern medical technology, and poor enlistment of community support.

The home hospital module offers most of the same medical components that are standard of care in an acute care hospital. The typical staff (medical doctor [MD], registered nurse [RN], case manager), diagnostics (blood tests, vital signs, telemetry, x-ray, and ultrasound), intravenous therapy, and oxygen/nebulizer therapy will all be available for home hospital. Optional deployment of food services, home health aide, physical therapist, occupational therapist, and social worker will be tailored to patient need. Home hospital improves upon the components of a typical ward's standard of care in several ways:

* Point of care blood diagnostics (results at the bedside in <5 minutes);
* Minimally invasive continuous vital signs, telemetry, activity tracking, and sleep tracking;
* On-demand 24/7 clinician video visits;
* 4 to 1 patient to MD ratio, compared to typical 16 to 1;
* Ambulatory/portable infusion pumps that can be worn on the hip;
* Optional access to a personal home health aide

Should a matter be emergent (that is, requiring in-person assistance in less than 20 minutes), then 9-1-1 will be called and the patient will be returned to the hospital immediately. In previous iterations of home hospital this happens in about 2% of patients.

Clinical parameters measured will be at the discretion of the physician and nurse, who treat the participant following evidence-based practice guidelines, just as in the usual care setting. In addition, the investigators will be tracking a wide variety of measures of quality and safety, including some measures tailored to each primary diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Resides within 5-mile radius of emergency room
* English- or Spanish-speaker
* Can identify a potential caregiver who agrees to stay with patient for first 24 hours of admission. Caregiver must be competent to call care team if a problem is evident to her/him.
* This criterion may be waived for highly competent patients at the patient and clinician's discretion.
* >=18 years old
* Primary diagnosis of cellulitis, heart failure, complicated urinary tract infection, or pneumonia that requires inpatient admission as determined by blinded emergency room team.

Exclusion Criteria:

* Undomiciled
* No working heat (October-April), no working air conditioning if forecast > 80°F (June-September), or no running water
* On methadone requiring daily pickup of medication
* In police custody
* Resides in facility that provides on-site medical care (e.g., skilled nursing facility)
* Domestic violence screen positive
* Cared for by a private primary care physician who rounds in the hospital
* Cannot establish peripheral access in emergency department (or access requires ultrasound guidance)
* Secondary condition: active non-melanoma/prostate cancer, end-stage renal disease, acute myocardial infarction, acute cerebral vascular accident, acute hemorrhage
* Primary diagnosis requires narcotics for pain control
* Cannot independently ambulate to bedside commode
* As deemed by on-call medical doctor, patient likely to require any of the following procedures: computed tomography, magnetic resonance imaging, endoscopic procedure, blood transfusion, cardiac stress test, or surgery
* For pneumonia:
* Most recent CURB65 > 3: new confusion, blood urea nitrogen > 19mg/dL, respiratory rate>=30/min, systolic blood pressure<90mmHg, Age>=65
* Most recent SMRTCO > 2: systolic blood pressure < 90mmHg (2pts), multilobar chest xray involvement (1pt), respiratory rate >= 30/min, heart rate >= 125, new confusion, oxygen saturation <= 90%
* Absence of clear infiltrate on imaging
* Cavitary lesion on imaging
* O2 saturation < 90% despite 5L O2
* For heart failure:
* Has a left ventricular assist device or paced rhythm
* Get with the Guidelines - Heart Failure (>10% in-hospital mortality) or The Acute Decompensated Heart Failure National Registry score (high risk or intermediate risk 1)
* Anasarca
* Pulmonary hypertension
* For complicated urinary tract infection:
* Absence of pyuria
* Most recent quick sepsis related organ failure assessment > 1
* Home hospital census is full (maximum 4 patients at any time)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total cost of hospitalization, $ | Day of admission to day of discharge

SECONDARY OUTCOMES:
Direct margin, $ | Day of admission to day of discharge
  Direct margin from total cost of hospitalization
Direct margin, modeled with backfill, $ | Day of admission to day of discharge
  Backfill uses a model that estimates the cost of patients who take the place of home hospital patients
Length of stay, days | Day of admission to day of discharge
Imaging, # | Day of admission to day of discharge
Lab Orders, # | Day of admission to day of discharge
Discharge Disposition | Day of discharge
  Routine, skilled nursing facility, home health, other
Readmission(s) after index hospitalization, y/n | Day of discharge to 30 days later
  Dichotomous outcome
Time to readmission after index hospitalization, days | Day of discharge to 30 days later
  Survival curve (hazard analysis)
Emergency Department (ED) observation stay(s) after index hospitalization, y/n | Day of discharge to 30 days later
  Dichotomous outcome
Time to ED observation stay(s) after index hospitalization, days | Day of discharge to 30 days later
  Survival curve (hazard analysis)
ED visit(s) after index hospitalization, y/n | Day of discharge to 30 days later
  Dichotomous outcome
Time to ED visit(s) after index hospitalization, days | Day of discharge to 30 days later
  Survival curve (hazard analysis)
Delirium, y/n | Day of admission to day of discharge
Transfer back to hospital, y/n | Day of admission to day of discharge
  intervention arm only
Hours of sleep, # | Day of admission to day of discharge
Daily steps, # | Day of admission to day of discharge
EuroQol -5D-5L, composite score | At admission, at discharge, and at 30 days after discharge
Short Form 1 | 30 days prior to admission (asked on day of admission), at admission, at discharge, and at 30 days after discharge
  1-5 Likert scale
Activities of daily living, score | 30 days prior to admission (asked on day of admission), at admission, at discharge, and at 30 days after discharge
Instrumental activities of daily living, score | 30 days prior to admission (asked on day of admission), at admission, at discharge, and at 30 days after discharge
3-item Care Transition Measure, score | 30 days after discharge
Picker Experience Questionnaire, score | 30 days after discharge
Global satisfaction with care, score | 30 days after discharge
Qualitative interview | 30 days after discharge

OTHER OUTCOMES:
Total cost of episode of care, $ | Day of admission to 30 days after discharge
  Exploratory; Subset of sample for which claims data is available
Intraveneous medications, days | Day of admission to day of discharge
  Exploratory
Intraveneous fluids, days | Day of admission to day of discharge
  Exploratory
Intraveneous diuretics, days | Day of admission to day of discharge
  Exploratory
Intraveneous antibiotics, days | Day of admission to day of discharge
  Exploratory
Supplemental oxygen required, days | Day of admission to day of discharge
  Exploratory
Nebulizer treatment, days | Day of admission to day of discharge
  Exploratory
Medical Doctor sessions, # notes | Day of admission to day of discharge
  Exploratory
Consultant sessions, # notes | Day of admission to day of discharge
  Exploratory
Physical therapy/occupational therapy sessions, # notes | Day of admission to day of discharge
  Exploratory
Primary care provider follow-up within 14 days, y/n | Day of discharge to 14 days later
  Exploratory
Skilled nursing facility utilization, days | Day of discharge to 30 days later
  Exploratory
Home health utilization, days | Day of discharge to 30 days later
  Exploratory
Fall, y/n | Day of admission to day of discharge
  Exploratory
Diagnosis of hospital-acquired or post-discharge deep vein thrombosis or pulmonary embolism | Day of admission to 30 days after discharge
  Exploratory
Hospital-acquired pressure ulcer, y/n | Day of admission to day of discharge
  Exploratory
Thrombophlebitis at peripheral intravenous site, y/n | Day of admission to day of discharge
  Exploratory
Catheter-associated urinary tract infection, y/n | Day of admission to day of discharge
  Exploratory
Clostridium difficile infection, y/n | Day of admission to day of discharge
  Exploratory
Methicillin resistant staph aureus infection, y/n | Day of admission to day of discharge
  Exploratory
Mortality during admission, y/n | Day of admission to day of discharge
  Exploratory
Post-discharge mortality, y/n | Day of discharge to 30 days later
  Exploratory
New arrhythmia, y/n | Day of admission to day of discharge
  Heart failure patients only; Exploratory
Hypokalemia, y/n | Day of admission to day of discharge
  Heart failure patients only; Exploratory
Acute kidney injury, y/n | Day of admission to day of discharge
  Heart failure patients only; Exploratory
Mean Likert scale pain score, 0-10 | Day of admission to day of discharge
  Exploratory
Pneumococcal vaccination if appropriate, y/n | Day of admission to day of discharge
  Pneumonia patients only; Exploratory
Influenza vaccination if appropriate, y/n | Day of admission to day of discharge
  Pneumonia patients only; Exploratory
Smoking cessation counseling if appropriate, y/n | Day of admission to day of discharge
  Pneumonia and heart failure patients only; Exploratory
Evaluation of ejection fraction as assessed by echocardiogram or other appropriate study, scheduled or completed, if not done within 1 year; y/n | Day of admission to day of discharge
  Heart failure patients only; Exploratory; appropriate studies include cardiac magnetic resonance imaging, radionuclide ventriculography, single photon emission computed tomography myocardial perfusion imaging, or left ventriculography
Angiotensin converting enzyme inhibitor or angiotensin receptor blocker for heart failure with reduced ejection fraction (ejection fraction < 40%), y/n | Day of admission to day of discharge
  Heart failure patients only; Exploratory
Beta blocker for heart failure with reduced ejection fraction (ejection fraction < 40%), y/n | Day of admission to day of discharge
  Heart failure patients only; Exploratory
Aldosterone antagonist for heart failure with reduced ejection fraction (ejection fraction < 40%), y/n | Day of admission to day of discharge
  Heart failure patients only; Exploratory
Lipid lowering for coronary artery disease, peripheral vascular disease, cerebrovascular accident, or diabetes, y/n | Day of admission to day of discharge
  Heart failure patients only; Exploratory
Smoking status post-discharge | 30 days after day of discharge
  Heart failure and pneumonia patients only; Exploratory; current/never/quit.
Use of inappropriate medications in the elderly, y/n | Day of admission to day of discharge
  Exploratory; using Screening Tool of Older Persons' potentially inappropriate Prescriptions (STOPP) and Beers criteria
Use of Foley catheter, y/n | Day of admission to day of discharge
  Exploratory
Use of restraints, y/n | Day of admission to day of discharge
  Exploratory
>3 medications added to medication list, y/n | Day of discharge (compared with preadmission med list)
  Exploratory
Patient health questionnaire-2, score | 30 days prior to admission (asked on day of admission), at admission, at discharge, and at 30 days after discharge
  Exploratory
Patient-Reported Outcomes Measurement Information System Emotional Support Short Form 4a, score | 30 days prior to admission (asked on day of admission), at admission, at discharge, and at 30 days after discharge
  Exploratory
Walk around ward/home, y/n | Day of discharge
  Exploratory
Get to (non-commode) bathroom, y/n | Day of discharge
  Exploratory
Walk 1 flight of stairs, y/n | Day of discharge
  Exploratory
Visit with friends/family, y/n | Day of admission to day of discharge
  Exploratory
Walk outside around my home, y/n | 30 days after discharge
  Exploratory
Go shopping, y/n | 30 days after discharge
  Exploratory
Time from admission decision to assessment by research assistant, minutes | Day of admission
  Exploratory
Time from research assistant assessment to emergency department dismissal, minutes | Day of admission
  Exploratory
Time from arrival home or to floor and medical doctor evaluation, minutes | Day of admission
  Exploratory
Time from arrival home or to floor and registered nurse evaluation, minutes | Day of admission
  Exploratory
Average Registered nurse to patient ratio | Day of admission to day of discharge
  Exploratory
Number of registered nurse visits, total | Day of admission to day of discharge
  Exploratory
Number of "on call" medical doctor interactions (video or phone), total | Day of admission to day of discharge
  Exploratory, intervention arm only
Number of "on call" medical doctor in-person visits, total | Day of admission to day of discharge
  Exploratory, intervention arm only
Duration of 1st registered nurse visit, minutes | Day of admission
  Exploratory, intervention arm only
Average Duration of subsequent registered nurse visit, minutes | Day of admission to day of discharge
  Exploratory, intervention arm only

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Schnipper, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leff B, Burton L, Mader SL, Naughton B, Burl J, Inouye SK, Greenough WB 3rd, Guido S, Langston C, Frick KD, Steinwachs D, Burton JR. Hospital at home: feasibility and outcomes of a program to provide hospital-level care at home for acutely ill older patients. Ann Intern Med. 2005 Dec 6;143(11):798-808. doi: 10.7326/0003-4819-143-11-200512060-00008. PMID 16330791
- [Background] Cryer L, Shannon SB, Van Amsterdam M, Leff B. Costs for 'hospital at home' patients were 19 percent lower, with equal or better outcomes compared to similar inpatients. Health Aff (Millwood). 2012 Jun;31(6):1237-43. doi: 10.1377/hlthaff.2011.1132. PMID 22665835
- [Background] Hung WW, Ross JS, Farber J, Siu AL. Evaluation of the Mobile Acute Care of the Elderly (MACE) service. JAMA Intern Med. 2013 Jun 10;173(11):990-6. doi: 10.1001/jamainternmed.2013.478. PMID 23608775
- [Background] Fong TG, Tulebaev SR, Inouye SK. Delirium in elderly adults: diagnosis, prevention and treatment. Nat Rev Neurol. 2009 Apr;5(4):210-20. doi: 10.1038/nrneurol.2009.24. PMID 19347026
- [Background] Counsell SR, Holder CM, Liebenauer LL, Palmer RM, Fortinsky RH, Kresevic DM, Quinn LM, Allen KR, Covinsky KE, Landefeld CS. Effects of a multicomponent intervention on functional outcomes and process of care in hospitalized older patients: a randomized controlled trial of Acute Care for Elders (ACE) in a community hospital. J Am Geriatr Soc. 2000 Dec;48(12):1572-81. doi: 10.1111/j.1532-5415.2000.tb03866.x. PMID 11129745
- [Background] Montalto M. The 500-bed hospital that isn't there: the Victorian Department of Health review of the Hospital in the Home program. Med J Aust. 2010 Nov 15;193(10):598-601. doi: 10.5694/j.1326-5377.2010.tb04070.x. PMID 21077817
- [Derived] Levine DM, Ouchi K, Blanchfield B, Diamond K, Licurse A, Pu CT, Schnipper JL. Hospital-Level Care at Home for Acutely Ill Adults: a Pilot Randomized Controlled Trial. J Gen Intern Med. 2018 May;33(5):729-736. doi: 10.1007/s11606-018-4307-z. Epub 2018 Feb 6. PMID 29411238